CLINICAL TRIAL: NCT05455918
Title: Non-randomized, Phase II, Open-label Study for Efficacy and Safety of Consolidation Paclitaxel/Ifosfamide/Cisplatin (TIP) Chemotherapy for High Risk Pediatric Germ Cell Tumor
Brief Title: Paclitaxel/Ifosfamide/Cisplatin Chemotherapy for High Risk Pediatric Germ Cell Tumor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0658
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Pediatric Germ Cell Tumor
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIP treatment arm (Experimental)
  Interventions: Drug: TIP treatment (paclitaxel/ifosfamide/cisplatin)

INTERVENTIONS:
Drug: TIP treatment (paclitaxel/ifosfamide/cisplatin) — Paclitaxel 240mg/m2/day D1 (total 240mg/m2) Ifosfamide 1.5g/m2/day D2~5 (total 6g/m2) Cisplatin 25mg/m2/day D2~5 (total 100mg/m2)

SUMMARY:
Germ cell tumor has generally good prognosis, but high risk germ cell tumor has still very poor prognosis. There remains the need of further improvement with other chemotherapy strategy. Especially more than 11 years old, mediastinal germ cell tumor, stage 3 or 4 extragonodal germ cell tumor or the remained tumor after the primary treatment are the group with the poorest prognosis.

Paclitaxel is widely used chemotherapeutic agent in adults and the experience of the agent has also been accumulated in children. The paclitaxel, ifosfamide, cisplatin (TIP) regimen has been used 2nd-line treatment for germ cell tumor and there is some promising result of the role of TIP in first line germ cell tumor treatment. In high risk pediatric germ cell tumor patients, TIP regimen will be able to reduce lung toxicity from the bleomycin as the standard regimen and to improve the survival. In this trial, the efficacy and safety of TIP as the first line treatment for germ cell tumor will be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Over 1 year old and less than 20 years old
* Pathologically or cytologically diagnosed germ cell tumor
* Germ cell tumor which has not been treated previously
* Higher than stage II (stage I should be excluded)
* Pathologic type

  1. embryonal carcinoma
  2. choriocarcinoma
  3. yolk sac tumor
  4. teratoma with malignant germ cell tumor elements
* High risk definition

  1. More than 11 years old, male or female
  2. Less than 11 years old, male or female

     1. Extragonodal germ cell tumor, stage III
     2. Extragonodal germ cell tumor, stage IV
     3. Ovarian germ cell tumor, stage IV
* More than 8 weeks of life expectancy
* performance level : ECOG Performance score 0, 1, or 2
* informed consent should be obtained

Exclusion Criteria:

* pregnancy or lactating patients (fertile men or women should agree to avoid pregnancy during the trial period)
* previously reported allergy or hypersensitivity to trial chemotherapeutic agent
* severe hypersensitivity to the agent containing Cremophor R EL (polyoxyethylated castor oil)
* Acceptable organ functions

  1. Bone marrow : Absolute neutrophil count >=1000/µL , platelet >= 100000/µL
  2. Renal function : serum creatinine ≤ 1.5 x upper limit of normal (ULN)
  3. Hepatic function : total bilirubin ≤ 1.5 x ULN, ALT ≤ 3.0 x UNL
  4. Cardiac Function : Ejection fraction ≥ 50%
  5. Uncontrolled infection
  6. Uncontrolled urinary obstruction
  7. Uncontrolled cystitis
* Followings will be excluded

  1. Mature teratoma
  2. Gliomatosis Peritonei
  3. Low Risk Germ Cell Tumor
  4. testicular stage I
  5. ovarian stage I
  6. recurrent, refractory tumor
* Concomitant other trial agent beside the agents in this trial
* Concomitant chemotherapeutic agents besides the agents in this trial

  1. Concomitant tumor other than germ cell tumor
  2. Other trial agents
  3. Other chemotherapeutic agents

Ages: 1 Year to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-07-26 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | 12weeks

SECONDARY OUTCOMES:
Overall Response Rate | 12 weeks and 18 weeks
Complete Response Rate | 18 weeks
Overall Survival | 3 years
Event Free Survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jung Woo Han, Principal Investigator — Department of Pediatric Hematology and Oncology, Yonsei Cancer Center, Yonsei University Health System.
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No